CLINICAL TRIAL: NCT06582771
Title: A Phase 2 Study of First-line Sotorasib for Patients With Advanced KRAS G12C-mutant Non-small Cell Lung Cancer
Brief Title: A Study of Sotorasib in People With Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-049
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non Small Lung Cancer
Keywords: Sotorasib; advanced KRAS G12C-mutant; 24-049
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Intervention Model Description: This will be a phase 2 study with a single cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sotorasib (Experimental): All patients will start at sotorasib 960 mg (8 pills) daily within 7 days of completion of the pretreatment tumor biopsy.
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Sotorasib 960 mg (8 pills) daily

SUMMARY:
The researchers are doing this study to see if sotorasib is a safe and effective treatment for people with advanced non-small cell lung cancer (NSCLC) with a KRAS G12C mutation who have not received treatment for their cancer since it became advanced. (Participants have not received a "first-line therapy" since their cancer became advanced.)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Biopsy-proven metastatic or recurrent non-small cell lung cancer
* KRAS G12C mutation on prior tumor biopsy or cell-free DNA (cfDNA) testing
* No prior therapy in the advanced setting
* Measurable disease per RECIST 1.1
* Karnofsky performance status (KPS) ≥ 70%
* Age ≥ 18
* Adequate organ function

  * Hemoglobin ≥ 9^9 g/dL
  * Platelets ≥ 75 x 10^9/L
  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L
  * AST < 3 x ULN (if liver metastases are present, < 5 x ULN)
  * ALT < 3 x ULN (if liver metastases are present, < 5 x ULN)
  * Alkaline phosphatase < 2 x ULN (if liver or bone metastases are present,< 3 xULN)
  * Total bilirubin ≤1.5 x ULN; subjects with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits
  * Serum creatinine < 1.5 x ULN or if available, calculated or measured creatinine clearance > 30 mL/min/1.73 m^2

In addition, patients must:

* Be willing to undergo pre-treatment and day 7-21 on-treatment tumor biopsies
* Decline first-line chemotherapy and/or anti-PD-(L)1 therapy, or previously have experienced disease progression after adjuvant or consolidation chemotherapy or anti-PD-(L)1 therapy for early stage (I-III) NSCLC

Before enrollment, a woman must be either:

* Not of childbearing potential: premenarchal; postmenopausal (>45 years of age with amenorrhea for at least 12 months); post-hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* Of childbearing potential and practicing effective method(s) of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies, as described below:

  * Practicing true abstinence (when this is in line with the preferred and usual lifestyle of the subject), which is defined as refraining from heterosexual intercourse during the entire period of the study, including up to 6 months after the last dose of study drug is given. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not consider an acceptable contraceptive method
* Have a sole partner who is vasectomized
* Practicing 2 methods of contraception, including one highly effective method (i.e., established use of oral, injected or implanted hormonal methods of contraception; placement of intrauterine device [IUD] or intrauterine system [IUS], AND, a second method (e.g., condom with spermicidal foam/gel/film/cream/suppository or collusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/ cream/suppository) Subjects must agree to continue contraception throughout the study and continuing through at least 7 days after the last dose of study drug
* NOTE: If the childbearing potential changes after start of the study (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) the woman must begin a highly effective method of birth control, as described above.
* A woman of childbearing potential must have a negative serum (b-human chorionic gonadotropin [b-hCG]) at Screening
* A man who is sexually active with a woman of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and his partner must also be practicing a highly effective method of contraception (i.e., established use of oral, injected or implanted hormonal methods of required to use contraception. The subject must also not donate sperm during the study and for at least 7 days after receiving the last dose of study drug.

contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]). If the subject is vasectomized, he must still use a condom (with or without spermicide), but his female partner is not required to use contraception. The subject must also not donate sperm during the study and for at least 7 days after receiving the last dose of study drug.

Exclusion Criteria:

* Symptomatic brain metastases
* Any radiotherapy within 1 week of starting treatment on protocol
* Any major surgery within 1 week of starting treatment on protocol
* Exposure to prior adjuvant or consolidation anti-PD-1 or PD-(L)1 therapy for stage I-III disease within 12 weeks of start of initiation of sotorasib
* Unresolved > grade 1 toxicity from any previous treatment
* Prior history of > grade 1 pneumonitis from any previous treatment
* Congestive heart failure defined as New York Heart Association (NYHA) Class III-IV or hospitalization for congestive heart failure (any NYHA class) within 6 months of study Day 1 Gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, uncontrolled inflammatory GI disease (eg, Crohn's disease, ulcerative colitis)
* Positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) o NOTE: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.

Positive hepatitis C antibody (anti-HCV)

o NOTE: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.

* Other clinically active or chronic liver disease
* Currently enrolled in another investigational device or drug study, or less than 28 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Use of known cytochrome P450 (CYP) 3A4 sensitive substrates (with a narrow therapeutic window), within 14 days or 5 half-lives (whichever is longer) of the drug or its major active metabolite, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator
* Use of strong inducers of CYP3A4 within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator
* Use of P-gp substrates within 14 days or 5 half-lives (whichever is longer) prior to study day 1 that was not reviewed and approved by the principal investigator
* Patients who do not agree to pre-treatment and on-treatment tumor biopsies during the informed consent process will be excluded from the study. Patients who agree to pre-treatment and on-treatment tumor biopsies, but in whom either biopsy is ultimately deemed unsafe by the investigators/treatment team, will be allowed to participate in the study and will remain evaluable for the clinical endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Response to therapy | within 6 month of therapy
  will be assessed with serial CT chest/abdomen/pelvis every 2 cycles (6 weeks), with response evaluated by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Riely, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm